CLINICAL TRIAL: NCT04463706
Title: Clinical Characterization of CoVid19 Infection: Prognostic Stratification and Complications
Brief Title: COVID19 Severity Prediction and Health Services Research Evaluation
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Hospital Costa del Sol (Other); Hospital del Mar (Other); University Hospital of the Nuestra Señora de Candelaria (Other); Instituto de Salud Carlos III (Other Government); Hospital Universitario Araba (Other); Biobizkaia Health Research Institute (Other Government); Hospital de Basurto (Other); Hospital Donostia (Other)
Responsible Party: Principal Investigator, Susana García Gutiérrez, PhD, Hospital Galdakao-Usansolo
Other Study IDs: COVID19_0459
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Covid19
Keywords: COVID; Risk stratification; Health services research; Cost-effectiveness; Equity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19 REDISSEC: Patients admitted (confirmed cases) by CoVid-19, excluding paediatric population. No losses are expected. A case of SARS-CoV-2 infection is defined as one that meets the laboratory criteria: PCR positive for a specific gene [RdRp or S gene] or PCR positive for at least 2 genes used for screening [E or N gene].
  Interventions: Other: Predictors adverse evolution
- COVID19 Basque Country: All people from thw Basque Country positive to CoVid-19. A case of SARS-CoV-2 infection is defined as one that meets the laboratory criteria: PCR positive for a specific gene [RdRp or S gene] or PCR positive for at least 2 genes used for screening [E or N gene], or, as well and in the general population of the Basque Country, by detection of COVID-19 IgM or IgG antibodies.
  Interventions: Other: Predictors of health care provide

INTERVENTIONS:
Other: Predictors adverse evolution — Predictors adverse evolution in all hospital participant admitted patients
  Groups: COVID19 REDISSEC
Other: Predictors of health care provide — Predictors of death, unequity, variability in process of care, cost in all COVID positive patients form the Basque Country
  Groups: COVID19 Basque Country

SUMMARY:
1. Objectives: 1.-To create risk stratification scales of poor evolution in patients infected by SARS-CoV-2. 2.-Evaluate the accessibility and equity that these patients have had in the different care processes, diagnostic and therapeutic procedures, with special interest in patients who came from residences, by age, gender or geographic origin.3.-Evaluate the effectiveness of different therapeutic schemes that have been used in this pandemic. 4.-Evaluate the effectiveness of different diagnostic tests used to predict the poor evolution of these patients 5.- Evaluate the real costs associated with the treatment of hospitalized patients with COVID-19 ; 2. Methods: Information will be recorded from electronic medical record: epidemiological data, onset of symptoms, comorbidities and their treatments, symptoms, analytical data, vital signs, tests performed, treatments during admission and evolution up to 3 months after discharge. Statistical analysis: The investigators will use classic survival models, logistic regression, generalized linear models and also analysis using artificial intelligence techniques . Health care costs are assessed. Applications for decision making will be derived as a product.

DETAILED DESCRIPTION:
Background: One of the fundamental problems of this epidemic is determined by the high percentage of SARS-CoV-2 infected patients who present rapid clinical deterioration that makes them need care in critical units. Identifying which factors are related to these more severe conditions would allow us to assess whether preventive or therapeutic measures can be put in place in advance or to better plan the services to be provided to these patients, either in this wave of the pandemic or in those that may occur in the future.

Objectives: This project aims to create stratification scales of the risk of poor evolution in patients infected by SARS-CoV-2, defined as the appearance of clinical deterioration, ARDS, sepsis, SRIS, septic shock or death. Additional goals are: 1.-Evaluate the accessibility and equity that these patients have had in the different care processes, diagnostic and therapeutic procedures, with special interest in patients who came from residences, by age, gender or geographic origin. 2.-Evaluate the effectiveness of different therapeutic schemes that have been used in this pandemic. 3.-Evaluate the effectiveness of different diagnostic tests used to predict the poor evolution of these patients 4.- Evaluate the real costs associated with the treatment of hospitalized patients with COVID-19.

Methods: The information will be extracted from the electronic medical record mostly, but will have to be done manually for certain fundamental parameters of prediction (clinical manifestations, date of onset of symptoms and duration of symptoms, and epidemiological history). Statistical analysis: Logistic regression/survival models/artificial intelligence algorithms will be created for the prediction of poor evolution of patients with CoVid-19.

Two samples are included: 1st.-All people SARS-CoV-2 positive from the Basque Country (around 380000 people) from March 2020 to January 2022; 2nd.-Patients admitted for COVID 19 in the centers participating in the study during the first wave of the pandemic, until May 31, will be included (in the case of the Basque Country, some of these patients will come from the population sample #1 described before). If there were new waves of a certain entity (more than 100 admissions in a month per center), this information would also be collected later. With the information the investigators have so far, the investigators see that the investigators would have between 6000-7000 to select. Later, patients from the autumn wave would be collected, if it were given, until the end of May 2021, due to greater temporal similarity with the first wave.

Sampling: 1st sample. - All people SARS-CoV-2 positive from the Basque Country from March 2020 to January 2022. 2nd sample. -The information to be reviewed from the medical record will be collected from the first wave of the pandemic between March-May 2020, where a random sampling will be carried out . For the second wave of autumn-winter of 2020-2021, a random sample of patients will also be collected, enough to meet the estimated sample size for this second wave. If not, the sample size will be completed with patients from the first wave.

VARIABLES: 1st sample. Sociodemographic, baseline comorbidities (including those of the Charlson Comobidity Index and based on ICD codes), baseline treatments (based on the Anatomical, Therapeutic, Chemical [ATC] classification system) [19]; vaccination status; dates of hospital admission and discharge and whether patients were admitted to an intensive care unit (ICU); and vital status. From those attended at any ED, we recorded vital signs (body temperature, blood pressure, heart rate and O2 saturation), gasometry, laboratory and chest X Ray image test, all from the unified electronic database.

2nd sample. -Exposure: 1.-Sociodemographic data: Age, gender, residence (yes / no), country of origin. 2.- Personal history: associated diseases; Basal treatments, etc. 3.-History of the disease 4.-Physical examination at home or AP. 5.-Hospital history: symptoms on arrival at the emergency department, vital signs, signs and physical examination, Laboratory tests, chest radiography pattern, CAT pattern, established treatments, ICU data.

Outcomes: 1st sample. -Hospital, ICU admission and death up to 90 days. 2nd sample. - Clinical impairment: Dyspnea at rest, Development of ARDS, sepsis, SIRS, shock, ICU admission, Death (date). Relief of symptoms, days until the absence of disease, death.

Follow-up: 1st sample. -Hospital, ICU admission and death up to 90 days. 2nd sample (6 months). Readmissions, New diagnoses, Complications, Biomarkers of fibrogenesis, Results of the diagnostic procedure (radiographs, MRI, CT), Death (with date and cause) Costs (index and 6 months income): Emergency or programmed admission; number of days of admission (in each of the Units / Plants / ICU / Emergencies); laboratory tests (number and type); number of days in which respiratory support was required; treatments used throughout the stay (drug, dose, dosage, duration); diagnostic procedures (radiographs, MRI, CT, etc.) performed during the study period; surgical procedures performed; external consultations (number and Service); day hospital (number and procedures); AP and home visits (related to COVID-19).

DATA COLLECTION METHODS: 1st sample: All data on patients in the care of our health service are held in a unified electronic database. Analysts retrieved previously described data for all SARS-CoV-2 infected patients during the study period. 2nd sample. Manual data extraction will be carried out by reviewers under the supervision of each PI per center. All the collected data will be entered in the RedCap database. Once the information is extracted, a common database will be created for subsequent analysis.

STATISTIC ANALYSIS. The study unit will be the patient. A descriptive analysis of the entire sample will be carried out. A univariate analysis will be performed to determine potential factors or variables related to the outcome variables of interest. In the multivariate analysis, different models will be carried out according to the dependent variable of interest. In the case of dichotomous dependent variables, logistic regression and Lasso models will be used. Statistical significance will be assumed when p <0.05 and all analyzes will be performed using SAS v9.4 and R statistical software. Also, the prediction of the variables will be evaluated individually by measuring the statistical correlation between each variable and the poor evolution; and collectively looking at the ability to predict the bad evolution from combinations, which will be obtained by generating Association Rules between variables from the underlying statistical relationships.

The analysis of the comparative effectiveness between the different treatment options that have been observed will be carried out by intention to treat. In addition to descriptive statistical techniques, a time-to-event (mortality) survival analysis will be performed using multivariate Cox proportional hazards regression, and a parametric survival analysis with the corresponding distribution (Weibull, etc.) together with an estimate. of average survival. For the evaluation of comparative effectiveness, propensity score techniques will be used to create comparable treatment groups by adjusting baseline covariates by inverse weighting of treatment probability. Additionally, and because it is foreseeable that there will be multiple treatment groups, the specific estimation procedure called generalized boosted models will be applied.

For the analysis of cost data, both for the analysis of associated variables and for a cost comparison objective, GLM regression techniques will be used with the type of distribution that best fits the data (using the Modified Park Test ), although preferably the gamma and logarithm family will be used as the link. The data will be analyzed with the Stata v14.2 program.

ETHICAL AND CONFIDENTIALITY ASPECTS. The project has been evaluated by the research commissions and the Research Ethics Committee with Medicines (CEIm), where it has been approved. The laws on personal data will be followed (RGPD 2018) All information will be treated in an absolutely confidential manner.

Expected results: A prognostic stratification tool based on predictive models of poor evolution in CoVid-19 infection: clinical deterioration and development of ARDS, SRS, sepsis, and/or septic shock and/or death. This tool will help guide the most appropriate clinical management of patients, mainly those with the most severe presentations that may require attention in critical care units. Additionally, purposes of this study are also to provide information on the variability and costs in the provision of health care that may have been given, both in the use of diagnostic tests and in the use of different therapeutic options and also in the results finally obtained. The investigators seek to identify problems in the accessibility of different groups (elderly, people in residences, by gender, higher level of comorbidities, immigrants ...), and that can help us identify problems in equity in access to health services.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID19 people in the Basque country
* Patients admitted (confirmed cases) by CoVid-19

Exclusion Criteria:

* Pediatric population (for objective #1 only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Positive COVID19 people in the Basque Country
  * Patients admitted by Covid-19 to hospitals in the Basque Country, from 01/02/2020 to 01/04/2020
Sampling Method: Non-Probability Sample
Enrollment: 380000 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical deterioration | Admission
  Clinical deterioration: Resting dyspnoea (Breathing rate > 30 breaths/minute) or 93% oxygen saturation at rest and partial pressure of arterial oxygen ; (PaO2) /Inspired fraction of O2 <300 mm Hg
  * Development of ARDS, sepsis, SIRS, shock
  * entry in ICU(date and days of stay)
  * Decease (date)

SECONDARY OUTCOMES:
Relief of symptoms | Admission
  Relief of symptoms (days), days until absence of disease (negative test), .
Mortality | 6 months
  Mortality
Complications at follow up | 6 months
  readmissions, clinical complications
Cost | Admission
  Economic cost

CONTACTS AND LOCATIONS:
Overall Officials: Susana Garcia-Gutierrez, PhD, Principal Investigator — Hospital Galdakao-Usansolo
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quintana JM, Larrea N, Menendez L, Legarreta MJ, Gascon M, Garcia-Asensio J, Espana PP; COVID-Health Basque Country Research Group. Effectiveness of drugs employed in the treatment of COVID-19: real-world evidence. Expert Rev Respir Med. 2025 May;19(5):493-498. doi: 10.1080/17476348.2025.2488966. Epub 2025 Apr 13. PMID 40186558
- [Derived] Espana PP, Bilbao-Gonzalez A, Larrea N, Castillo-Sintes I, Garcia-Gutierrez S, Portuondo J, Villanueva A, Uranga A, Legarreta MJ, Gascon M, Quintana JM; COVID-Health Basque Country Research Group. Impact of prior SARS-COV-2 infection and vaccination on COVID-19 hospital admission and mortality amongst nursing home residents. Aging Clin Exp Res. 2023 Aug;35(8):1771-1778. doi: 10.1007/s40520-023-02446-3. Epub 2023 May 30. PMID 37249860
- [Derived] Garcia-Gutierrez S, Esteban-Aizpiri C, Lafuente I, Barrio I, Quiros R, Quintana JM, Uranga A; COVID-REDISSEC Working Group. Machine learning-based model for prediction of clinical deterioration in hospitalized patients by COVID 19. Sci Rep. 2022 May 2;12(1):7097. doi: 10.1038/s41598-022-09771-z. PMID 35501359
- [Derived] Portuondo-Jimenez J, Bilbao-Gonzalez A, Tiscar-Gonzalez V, Garitano-Gutierrez I, Garcia-Gutierrez S, Martinez-Mejuto A, Santiago-Garin J, Arribas-Garcia S, Garcia-Asensio J, Chart-Pascual J, Zorrilla-Martinez I, Quintana-Lopez JM; COVID-19-Osakidetza Working group. Modelling the risk of hospital admission of lab confirmed SARS-CoV-2-infected patients in primary care: a population-based study. Intern Emerg Med. 2022 Jun;17(4):1211-1221. doi: 10.1007/s11739-022-02931-z. Epub 2022 Feb 10. PMID 35143022
- [Derived] Esteban C, Villanueva A, Garcia-Gutierrez S, Aramburu A, Gorordo I, Quintana JM, Working Group TC. COPD in SARS-CoV-2 pandemic. baseline characteristics related to hospital admissions. Expert Rev Respir Med. 2022 Apr;16(4):477-484. doi: 10.1080/17476348.2022.2031985. Epub 2022 Apr 6. PMID 35060833
- [Derived] Espana PP, Bilbao A, Garcia-Gutierrez S, Lafuente I, Anton-Ladislao A, Villanueva A, Uranga A, Legarreta MJ, Aguirre U, Quintana JM; COVID-19-Osakidetza Working group. Predictors of mortality of COVID-19 in the general population and nursing homes. Intern Emerg Med. 2021 Sep;16(6):1487-1496. doi: 10.1007/s11739-020-02594-8. Epub 2021 Jan 5. PMID 33400164